CLINICAL TRIAL: NCT05361564
Title: A Window of Opportunity Study for Investigating Drug Tolerant Persister (DTP) to Preoperative Brigatinib in Resectable Non-small Cell Lung Cancer (NSCLC) Harboring ALK Fusions.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0569-001
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; neo-adjuvant; ALK fusion; drug tolerant persister(DTP)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — brigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brigatinib (Experimental)
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — After 7-day lead-in 90mg/day, brigatinib 180mg/day from 4 to 10weeks(optimal duration: 6 weeks)

SUMMARY:
This study is single arm, open label, phase II trial for resectable ALK+ NSCLC. Eligible patients will receive brigatinib after 7-day lead-in 90mg from 4 to 10 weeks.

The objective of this study is as follows.

* Primary objective: To identify molecular mechanism of DTP causing innate drug resistance to neoadjuvant brigatinib in resectable NSCLC harboring ALK fusion by analyzing single cell RNA-seq.
* Secondary objectives:

  1. To assess the pathologic response rate to neoadjuvant treatment with Brigatinib
  2. To evaluate the clinical efficacy in resectable ALK-positive NSCLC patients treated with brigatinib induction therapy
  3. To evaluate the successful curative resection rate
  4. To evaluate the safety of brigatinib as neoadjuvant treatment in resectable ALK-rearranged NSCLC patients.
  5. To investigate the changes of ALK rearrangement and other hot spot mutations by GUARDANT LUNAR assay of circulating tumor DNA present in blood plasma immediately with serial sampling.
  6. To assess of variant allele frequencies between pre-treatment and post-treatment sampling by GUARDANT LUNAR assay
  7. To explore cell-free biomarkers that may be predictive of response or primary resistance to brigatinib neoadjuvant therapy

DETAILED DESCRIPTION:
This study is single arm, open label, phase II trial for resectable ALK+ NSCLC. Eligible patients will receive brigatinib after 7-day lead-in 90 mg from 4 to 10 weeks. The surgery with curative intent will be performed within 4 - 10 weeks after initiating brigatinib (optimal duration: 6 weeks). The surgery with curative intent represents more than sublobar resection with mediastinal lymph node dissection. Patients take it up to the day before surgery and can be allow stop up to 3 days before surgery by physician's discretion.

Post-operative adjuvant treatment will be conducted based on the treating physician's best medical judgement.

Brigatinib will be administered orally at a dose of 90 mg QD for the first 7 days. Patients who have tolerated the 90 mg starting dose on Days 1 through 7 will be expected to increase their dose to 180 mg QD beginning on Day 8 and continuously every day, with a 28-day study procedure execution cycle. The study drug shall be taken approximately at the same time of the day each day. It may be taken with or without food. Patients shall be instructed to swallow the tablets whole and not crush or chew them. Patients will take the dose with water (recommended 240 mL). If a dose of brigatinib is missed or vomiting occurs after taking a dose, do not administer an additional dose and take the next dose of brigatinib at the scheduled time.

The patient's daily dose of brigatinib should not be increased to 180 mg if any of the following adverse reactions are experienced during treatment at 90 mg QD:

* Interstitial lung disease (ILD)/pneumonitis (any grade).
* Symptomatic bradycardia (Grade 2 or greater).
* Grade 2 or higher visual disturbance.
* Any other Grade 3 or higher adverse reaction.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 20 years or older.
2. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
3. Female patients who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse

   Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or
   * Agree to completely abstain from heterosexual intercourse
4. Treatment-naïve stage I to IIIa non-small cell lung cancer according to the AJCC 8th edition and amenable to surgical resection.
5. Documented ALK rearrangement (VENTANA ALK (D5F3) CDx Assay or appropriate diagnostic method)
6. Brain magnetic resonance imaging (MRI) (or CT if contraindication to MRI) within the last 60 days showing no evidence of metastatic disease
7. Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0 or 1
8. Documentation that the patient is a candidate for surgical resection of their lung cancer by certified surgeon.
9. Measurable disease defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
10. Clinical laboratory values as specified below within 4 weeks before the first dose of study drug:

    * ALT/aspartate aminotransferase (AST) ≤2.5 × upper limit of normal (ULN); ≤5 × ULN is acceptable if liver metastases are present.
    * Total serum bilirubin ≤1.5 × ULN (<3.0 × ULN for patients with Gilbert syndrome).
    * Estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2, using the modification of diet in renal disease (MDRD) equationd) Serum lipase ≤1.5 × ULN.
    * Absolute neutrophil count ≥1.5 × 10^9/L.
    * Platelet count ≥75 × 10^9/L.
    * Hemoglobin ≥8 g/dL.
11. Ability to swallow oral medications

Exclusion Criteria:

1. Clinical stage IIIb or IIIc or distant metastases (including malignant pleural effusion) identified in CT, PET-CT, brain imaging or biopsy.
2. Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug.
3. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
4. Treatment with any investigational products within 4 weeks before the first dose of study drug
5. Had major surgery within 30 days of the first dose of brigatinib. Minor surgical procedures such as catheter placement or minimally invasive biopsies are allowed.
6. Have been diagnosed with another primary malignancy other than NSCLC, except for adequately treated nonmelanoma skin cancer or cervical cancer in situ; definitively treated nonmetastatic prostate cancer; or patients with another primary malignancy who are definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy.
7. Have symptomatic brain metastasis (parenchymal or leptomeningeal). Patients with asymptomatic brain metastasis or who have stable symptoms that did not require an increased dose of corticosteroids to control symptoms in the past 7 days before the first dose of brigatinib may be enrolled.
8. Have current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging). Patients with leptomeningeal disease and without cord compression are allowed.
9. Have significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

   * Myocardial infarction within 6 months before the first dose of brigatinib.
   * Unstable angina within 6 months before first dose of brigatinib.
   * Congestive heart failure within 6 months before first dose of brigatinib.
   * History of clinically significant atrial arrhythmia (including clinically significant bradyarrhythmia), as determined by the treating physician.
   * Any history of clinically significant ventricular arrhythmia.
   * Had a cerebrovascular accident or transient ischemic attack within 6 months before first dose of brigatinib.
10. Have uncontrolled hypertension. Patients with hypertension should be under treatment on study entry to control blood pressure.
11. Have a history or the presence at baseline of pulmonary interstitial disease, drug-related pneumonitis, or radiation pneumonitis.
12. Have an ongoing or active infection, including, but not limited to, the requirement for intravenous antibiotics.
13. Have a known history of HIV infection. Testing is not required in the absence of history.
14. Have malabsorption syndrome or other GI illness that could affect oral absorption of brigatinib.
15. Have a known or suspected hypersensitivity to brigatinib or its excipients.
16. Are pregnant, planning a pregnancy, or breastfeeding.
17. Have any condition or illness that, in the opinion of the investigator, would compromise patient safety or interfere with the evaluation of brigatinib.
18. Received systemic treatment with strong cytochrome P-450 (CYP)3A inhibitors, strong CYP3A inducers, or moderate CYP3A inducers within 14 days before enrollment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
molecular candidates identified by analyzing scRNA-seq | 10weeks (after surgery)
  Molecular candidates identified by analyzing scRNA-seq from pre-treatment tumor biopsy specimens and tumor tissue acquired at the time of surgical resection.

SECONDARY OUTCOMES:
Pathologic complete response rate (pCR) | 10weeks (after surgery)
  absence of (0%) viable tumor present histologically in the resected tumor specimen
Major pathologic response (MPR) | 10weeks (after surgery)
  ≤10% residual viable tumor following neoadjuvant therapy
Disease-free survival (DFS) | Up to 2 years
Event free survival (EFS) | Up to 2 years
Overall survival (OS) | 6months
Overall survival (OS) | Up to 2 years
Objective response rate (ORR) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  CR+PR rate based on RECIST ver 1.1 criteria.
Rate of inability to undergo surgical resection | 10 weeks
Rate of conversion from operable to non-operative | 10weeks
  It will be recorded as rate of patients initially assessed as surgically resectable, who are subsequently unable to undergo surgical resection due to either treatment-related adverse events (AEs) or disease progression
Rate of surgical complications occurring post op period | 16weeks (6 weeks after surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No